CLINICAL TRIAL: NCT01776619
Title: A Double Blind (3rd Party Open) Randomized, Dose Escalation Study to Investigate the Safety, Tolerability, Pharmacokinetics of Repeat Doses PF-06305591 Combined With a Cross-over Relative Bioavailability and Food Effect Evaluation After Single Dose of PF-06305591 in Healthy Young Subjects
Brief Title: Safety and Tolerability Study of Multiple Doses of PF-06305591
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B5281002
Record Dates: First submitted 2013-01-23; First posted 2013-01-28 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-12

CONDITIONS: Healthy
Keywords: Safety; tolerability; PK

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Multiple Dose: Cohort 1 (Experimental)
  Interventions: Drug: PF-06305591; Drug: Placebo
- Multiple Dose: Cohort 2 (Experimental)
  Interventions: Drug: PF-06305591; Drug: Placebo
- Multiple Dose: Cohort 3 (Experimental)
  Interventions: Drug: PF-06305591; Drug: Placebo
- Multiple Dose: Cohort 4 (Experimental)
  Interventions: Drug: PF-06305591
- Relative Bioavilability: Cohort 1 (Experimental)
  Interventions: Drug: PF-06305591

INTERVENTIONS:
Drug: PF-06305591 — 14 day repeated 20mg BID doses
  Arms: Multiple Dose: Cohort 1
Drug: Placebo — 14 day repeated BID doses
  Arms: Multiple Dose: Cohort 1
Drug: PF-06305591 — 14 day repeated 80mg BID doses
  Arms: Multiple Dose: Cohort 2
Drug: Placebo — 14 day repeated BID doses
  Arms: Multiple Dose: Cohort 2
Drug: PF-06305591 — 14 day repeated 40mg BID doses
  Arms: Multiple Dose: Cohort 3
Drug: Placebo — 14 day repeated BID doses
  Arms: Multiple Dose: Cohort 3
Drug: PF-06305591 — 14 day repeated BID doses
  Arms: Multiple Dose: Cohort 4
Drug: PF-06305591 — relative bioavailability tablet vs. solution and food effect at 50mg dose
  Arms: Relative Bioavilability: Cohort 1

SUMMARY:
Safety, tolerability and PK of repeated doses of PF-06305591 will be evaluated in young healthy volunteers toghether with food effect on relative bioavailability of solid formulation after single dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects of non childbearing potential, between the ages of 21 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG and clinical laboratory tests

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy).

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2013-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | 14 days
  Counts of participants who had treatment-emergent adverse events (TEAEs), defined as newly occurring or worsening after first dose. Relatedness to [study drug] was assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category were counted once within the category.
Maximum Observed Plasma Concentration (Cmax) | 14 days
Area under the Concentration-Time Curve (AUC) | 14 days
  AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption.
Area Under the Curve from Time Zero to end of dosing interval (AUCtau) | 14 days
  AUC is a measure of the serum concentration of the drug over time interval. It is used to characterize drug absorption.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B5281002&StudyName=Safety%20and%20Tolerability%20Study%20of%20Multiple%20Doses%20of%20PF-06305591